CLINICAL TRIAL: NCT06947421
Title: Effectiveness of McKenzie and Standard Neck Exercises on Craniovertebral Angle, Hand Grip Strength, and Psychosocial Status in Individuals With Forward Head Posture- Randomized Assessor Blinded Clinical Trial
Brief Title: The Effect of Different Exercises on Craniovertebral Angle in Individuals With Forward Head Posture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Esra BECENI, lecturer, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2206
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Forward Head Posture
Keywords: forward head posture; craniovertebral angle; McKenzie; Standard Neck Exercises

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, assessor-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization will be done by the sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Exercise Group (MG) (Experimental): Participants in this group will follow a McKenzie-based cervical exercise program consisting of four specific movements: retraction, rotation, lateral flexion, and combined rotation.
  Interventions: Behavioral: McKenzie Exercise
- Standard Neck Exercise Group (SG) (Experimental): Participants in this group will follow a standard cervical postural correction program focused on strengthening deep cervical flexors and scapular retractors, and stretching cervical extensors and pectoralis muscles.
  Interventions: Behavioral: Standard Neck Exercise

INTERVENTIONS:
Behavioral: McKenzie Exercise — Exercises will be performed in seated or supine positions, 15 repetitions per session, twice daily, for a total duration of 6 weeks. The program will begin with physiotherapist-supervised sessions and continue at home with guidance via a digital training manual. Weekly follow-up and progress will be ensured through individual exercise diaries. Participants missing two consecutive days of exercise will be excluded from the study. Includes:
  * Cervical retraction in sitting and supine positions
  * Cervical rotation to both sides
  * Lateral flexion of the neck
  * Combined chin rotation toward the shoulder
  Arms: McKenzie Exercise Group (MG)
Behavioral: Standard Neck Exercise — The protocol includes chin tucks, chin drop stretches, scapular retraction with resistance, and both unilateral and bilateral pectoral stretching. Exercises will be performed twice daily, 15 repetitions per session, over a period of 6 weeks. Exercise progression will be adapted biweekly based on participant tolerance. Includes:
  * Chin tucks in supine with progressive hold durations
  * Chin drop stretch in sitting with optional manual assistance
  * Scapular retraction using theraband or weights
  * Pectoral muscle stretching using doorway and seated techniques
  Arms: Standard Neck Exercise Group (SG)

SUMMARY:
Forward head posture (FHP) is a prevalent postural misalignment commonly attributed to prolonged exposure to poor ergonomic conditions and insufficient physical activity. This condition adversely affects craniovertebral angle (CVA), cervical muscle activity, and upper extremity function, ultimately compromising overall physical health and quality of life. Current literature highlights the corrective effects of McKenzie exercises on postural awareness and cervical alignment, while standard neck exercises are frequently employed to address muscular imbalances and alleviate posture-related pain and functional limitations. However, studies that directly compare these two exercise approaches in individuals with FHP particularly in terms of their short-term effects on craniovertebral angle, hand grip strength, and psychosocial outcomes remain scarce. Accordingly, the present study aims to fill this critical gap by conducting a multidimensional analysis of the immediate effects of McKenzie versus standard neck exercise programs in individuals with FHP, thereby contributing meaningful insights to clinical rehabilitation practices.

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common postural misalignment characterized by the anterior positioning of the head relative to the trunk in the sagittal plane. It is frequently associated with poor ergonomic habits, prolonged screen time, heavy backpack use, and lack of physical activity. This postural deviation can lead to upper cervical hyperextension, lower cervical and upper thoracic flexion, increased muscle tension, and long-term dysfunctions in the musculoskeletal, neurological, and vascular systems.

The craniovertebral angle (CVA) is a commonly used and reliable method for evaluating FHP. A CVA less than 50 degrees is considered indicative of forward head posture. Current literature supports the use of exercise interventions to improve CVA and reduce the symptoms associated with postural abnormalities.

The McKenzie method is based on directional preference and repetitive movements, aiming to enhance postural awareness and spinal alignment. Standard neck exercises, frequently used in clinical practice, aim to improve muscular balance, cervical alignment, and reduce neck pain.

Although both exercise methods have shown individual effectiveness in improving posture and function, few studies have directly compared their effects on both structural and functional outcomes. Additionally, hand grip strength and psychosocial factors are often overlooked, despite their importance in evaluating upper extremity function and overall well-being in individuals with FHP.

This randomized, assessor-blinded clinical trial aims to compare the short-term effects of McKenzie exercises and standard neck exercises on craniovertebral angle, hand grip strength, and psychosocial status in individuals with forward head posture. The results will contribute to clinical knowledge regarding effective rehabilitation strategies for postural dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with forward head posture, defined by a craniovertebral angle (CVA) of less than 50°, based on established diagnostic criteria
* Age between 18 and 30 years
* Pain intensity greater than 3 on the Visual Analog Scale (VAS)
* Mild to moderate neck disability, indicated by a Neck Disability Index (NDI) score below 15 out of 50
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Presence of medical contraindications to exercise
* Regular engagement in structured spinal exercise programs
* History of spinal surgery
* Diagnosis of cancer or other malignant conditions
* Presence of an implanted cardiac pacemaker
* Visual, auditory, or cognitive impairments that would prevent adherence to the exercise protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
1.Craniovertebral Angle (CVA) | through study completion, an average of 6 months
  CVA is used to assess forward head posture. Participants will be asked to stand in a natural and relaxed posture while focusing on a marked point at eye level on the wall. A lateral photograph will be taken using a Iphone 13 camera mounted on a tripod at shoulder height and placed 1.5 meters from the participant. The spinous process of the C7 vertebra and the tragus of the ear will be marked. The angle between the line connecting the tragus to C7 and a horizontal reference line will be calculated using the ImageJ software. The measurement results will be recorded on the evaluation form.
  Analysis Metric: Change in CVA (degrees)

SECONDARY OUTCOMES:
2.Cognitive Exercise Therapy Approach Scale (BETY) | through study completion, an average of 6 months
  The BETY scale will be used to assess participants' biopsychosocial status, including emotional state, functionality, fatigue, pain, sleep quality, and social/sexual life. The scale consists of 30 items scored on a 0-4 Likert scale, with a total score range of 0-120. Higher scores indicate greater biopsychosocial impairment.
  Analysis Metric: Total score (0-120)
3.Hand Grip Strength (HGS) | through study completion, an average of 6 months
  Grip strength will be measured using a Baseline hydraulic hand dynamometer. Participants will be seated or standing upright with the shoulder in adduction, elbow at 90° flexion, wrist in 0-30° extension and 0-5° ulnar deviation. They will be instructed to squeeze the dynamometer with maximum effort for 3 seconds. The test will be performed three times for each hand (starting with the dominant hand), and the highest value from each will be recorded.
  Analysis Metric: Maximum grip strength in kilograms (kg)
4.Neck Disability Index (NDI) | through study completion, an average of 6 months
  The Neck Disability Index is a standardized self-reported questionnaire used to assess the impact of neck pain on daily living activities. This scale evaluates the individual's functional status through self-assessment of neck pain, including domains such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreational activities. Each section is scored on a scale from 0 ("no pain") to 5 ("the worst pain imaginable"). The scores from each section are summed and expressed as a percentage to determine the overall level of disability. Interpretation categories are as follows: 0-8% = no disability, 10-28% = mild, 30-48% = moderate, 50-64% = severe, and 70-100% = complete disability
5. Visual Analog Scale (VAS) for Neck Pain | through study completion, an average of 6 months
  Cervical pain intensity will be assessed using a 10-cm horizontal VAS. Participants will mark their current level of pain on the line, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Analysis Metric: Pain score (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy; Esra Beceni, PhD Student, Principal Investigator — Bahcesehir University, Graduate Education Institute; Büşra Tamgüç, PhD Student, Study Chair — Bahcesehir University, Graduate Education Institute; Gülay Yalcin, PhD, Study Chair — Mudanya University, Faculty of Health Sciences, Department of Physiotherapy
Locations (1):
- Mudanya University, Bursa, Turkey (Türkiye)